CLINICAL TRIAL: NCT03012516
Title: Physical Activity on Prescription With Two Different Strategies. One Year Follow-up Regarding Physical Activity Level, Metabolic Health and Health-related Quality of Life. A Randomized Controlled Trial.
Brief Title: Physical Activity on Prescription in Patients With Metabolic Risk Factors.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAP-study RCT 206261
Record Dates: First submitted 2016-12-30; First posted 2017-01-06 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Health Behavior; Activities of Daily Living; Metabolic Syndrome X; Quality of Life
Keywords: Physical Therapy Specialty; Exercise Test; Prescriptions; Counseling; Primary Health Care; Exercise
MeSH Terms: conditions — Health Behavior; Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PAP-treatment by physiotherapist. (Experimental): Enhanced PAP-support by physiotherapist including fitness test, individualized dialogue concerning PA, prescribed PAP and a 7 times follow-up during the one year intervention..
  Interventions: Behavioral: PAP-treatment by physiotherapist
- Ordinary PAP-treatment at the health care centre. (Active Comparator): Ordinary PAP-treatment at the health care centre including individualized dialogue concerning PA, prescribed PAP and an individually adjusted follow-up.
  Interventions: Behavioral: Ordinary PAP-treatment at the health care center

INTERVENTIONS:
Behavioral: PAP-treatment by physiotherapist
  Arms: PAP-treatment by physiotherapist.
Behavioral: Ordinary PAP-treatment at the health care center
  Arms: Ordinary PAP-treatment at the health care centre.

SUMMARY:
The aim of this study is to evaluate a one year intervention with physical activity on prescription (PAP) treatment for patients in a primary health care center setting versus an enhanced PAP-support with physiotherapist regarding physical activity (PA) level, metabolic health effects and health-related quality of life.

One hundred ninety patients, 27-85 years, physically inactive, having at least one component of the metabolic syndrome and not responding with increased PA level after a 6-months PAP-treatment in primary health care centre are randomized to either enhanced support by physiotherapist (Intervention group) or continued ordinary PAP-treatment at the health care centre (Control group).

DETAILED DESCRIPTION:
Aim:

The aim is to evaluate whether an enhanced support with physiotherapist for patients who are non-responders to PAP-treatment at 6 months follow-up in a primary health care centre setting influences physical activity level, metabolic health effects and health-related quality of life.

Methods:

Study design:

This is a randomized controlled trial (RCT) with two arms: one intervention group and one control group. The present study is part of an ongoing study including 444 patients with a 5 years follow-up.

Study population:

The study population includes 190 patients, 27-85 years, having at least on component of the metabolic syndrome (metS) and non-responding to PAP-treatment initiated at health care centre. The patients randomizes to either enhanced PAP-support by physiotherapist (Intervention group n = 98) or continued ordinary PAP-treatment at the health care centre (Control group n = 92).

Intervention:

In the control group, PAP-treatment is offered by authorized personnel, mainly nurses and includes an individualized dialogue concerning PA, prescribed PAP and an individually adjusted follow-up. The intervention by physiotherapist includes fitness test using an ergometer bicycle. The result from the ergometer bicycle test forms the basis for a continuing motivating dialogue concerning physical activity and an individually dosed physical activity regarding frequence, duration and intensity with a prescribed PAP. The patient is supported by physiotherapist 7 times during the one year intervention.

Measurements:

For both groups, the patients PA-level, metabolic health and health related quality of life is measured at baseline and one-year follow-up, at the health care centre. In the intervention group, the ergometer bicycle test is conducted by the physiotherapist.

Statistical analysis:

The size of the study is calculated based on a power of 90%, to detect a difference of 20% in physical activity level between the intervention (40% responders) and control (20% responders) groups referred to physical activity level ≥5 points, at a significance level of 0.05. Intention-to-treat analysis will be used. Data will be processed using Paired samples t-test or Wilcoxon sign-rank test based on data level in within group analyses. Analyses between intervention and control group will be performed using Independent samples t-test or Mann Whitney U-test. Statistical significance is set at p ≤ 0.05.

Hypothesis:

An enhanced PAP-support by physiotherapist gives room for enlarged effects on physical activity level with an opportunity to influence cardiorespiratory fitness, metabolic health and health related quality of life.

Clinical implication:

An increased physical activity level in the non-responder group via an individually designed PAP-support by physiotherapist will increase the possibility to save time and resources for both the patients and health care system. Evaluating effects on cardiorespiratory fitness in addition to metabolic health and health related quality of life gives an immersed understanding of the health effects due to this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Physically inactive according to ACSM/AHA public health recommendation from 2007.
* Having at least one component of the metS present according to the NCEP classification.
* Receiving PAP-treatment.
* Understanding the Swedish language.

Exclusion Criteria:

* The patient decline to participate.

Ages: 27 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Change in self-assessed PA-level according to the public health recommendation. | Change between baseline and one year follow-up.
  Self-assessment of PA-level according to American college of sports medicine (ACSM) and American heart association (AHA) public health recommendation 2007. The patient responds to two PA questions, where 30 minutes of moderate-intensity PA per day results in 1 point and 20 minutes of more vigorous-intensity PA per day results in 1.7 point during each specific day of the week. A value of <5 points indicates an inadequate PA level.
Change in self-assessed PA-level - IPAQ | Change between baseline and one year follow-up.
  The International physical activity questionnaire (IPAQ) assessing the level of PA during the last seven days. The instrument is extensively tested and translated into Swedish and vigorous-, moderate-intensity PA, walking and sitting time can be assessed.
Change in self-assessed PA-level - SGPALS | Change between baseline and one year follow-up.
  The Saltin-Grimby physical activity level scale (SGPALS) assessing leisure time PA during the past year in four different levels, from sedentary/physically inactive to vigorous physically active. The levels has been validated against e.g. metabolic risk factors and has been published in an updated Swedish form.
Change in self-assessed PA-level - a six grade PA scale | Change between baseline and one year follow-up.
  A six-grade PA scale is a further development of the SGPALS (Frändin/Grimby), and includes household activities. This scale correlates with physical performance and self-assessed fitness and is used to classify PA among elderly

SECONDARY OUTCOMES:
Change in anthropometrics - Body mass index (BMI) | Change between baseline and one year follow-up.
  Body weight is measured with light clothing and without shoes to the nearest 0.1 kg using an electric scale (Carl Lidén AFW D300, Jönköping, Sweden). Body height is measured in an upright position without shoes to the nearest 0.5 cm using a scale fixed to the wall (Personmått PEM 136, Hultafors, Sweden) and BMI in kg/m^2 is calculated.
Change in anthropometrics - Waist circumference (WC) | Change between baseline and one year follow-up.
  WC, to the nearest 0.5 cm, is measured in a standing exhaled position, with a measuring-tape (Kirchner Wilhelm, Aspberg, Germany) placed on the patients skin between the lower rib and the iliac crest. The cut-off values of metS components according to The National Cholesterol Education Program (NCEP) classification includes WC > 88 cm for women, >102 cm for men.
Change in systolic blood pressure (SBP) | Change between baseline and one year follow-up.
  SBP is measured in mmHg according to guidelines, after 5 minutes rest, with the patient seated, having a blood pressure sphygmomanometer (Omron HEM-907, Kyoto, Japan) attached to the right upper arm at the level of the heart. The cut-off values of metS components according to The National Cholesterol Education Program (NCEP) classification includes SBP ≥ 130 mmHg
Change in diastolic blood pressure (DBP) | Change between baseline and one year follow-up.
  DBP is measured in mmHg according to guidelines, after 5 minutes rest, with the patient seated, having a blood pressure sphygmomanometer (Omron HEM-907, Kyoto, Japan) attached to the right upper arm at the level of the heart. The cut-off values of metS components according to The National Cholesterol Education Program (NCEP) classification includes DBP ≥ 85 mmHg
Change in blood samples - Plasma glucose after an overnight fast (FPG). | Change between baseline and one year follow-up.
  FPG measured in mmol/l and analyzed according to the European Accreditation system. The cut-off values of metS components according to The National Cholesterol Education Program (NCEP) classification includes FPG ≥ 6.1.
Change in blood samples - Triglycerides (TG). | Change between baseline and one year follow-up.
  TG measured in mmol/l and analyzed according to the European Accreditation system. The cut-off values of metS components according to The National Cholesterol Education Program (NCEP) classification includes TG ≥ 1.7 mmol/l.
Change in blood samples - Cholesterol. | Change between baseline and one year follow-up.
  Cholesterol measured in mmol/l and analyzed according to the European Accreditation system.
Change in blood samples - High Density Lipoprotein (HDL). | Change between baseline and one year follow-up.
  HDL measured in mmol/l and analyzed according to the European Accreditation system.The cut-off values of metS components according to The National Cholesterol Education Program (NCEP) classification includes HDL < 1.3 mmol/l for women, < 1.0 mmol/l for men.
Change in blood samples - Low Density Lipoprotein (LDL). | Change between baseline and one year follow-up.
  LDL measured in mmol/l and analyzed according to the European Accreditation system.
Change in health related quality of life - Short Form 36 (SF-36) | Change between baseline and one year follow-up.
  Assessed with the Swedish version of the Short Form 36 (SF-36 Standard Swedish Version 1.0) which includes 36 questions. It generates eight health concepts: physical functioning (PF), role physical functioning (RP), bodily pain (BP), general health (GH), vitality (VT), social function (SF), role emotional functioning (RE) and mental health (MH). The health concepts are converted to 0-100 points where higher values represents a better health-related quality of life. The different health concepts of SF-36 are also grouped into a physical component summary (PCS) and mental component summary (MCS) respectively. SF-36 has shown good to excellent internal consistency reliability and is validated in a representative sample of Swedish population.

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Cider, PhD, Principal Investigator — Department of Health and Rehabilitation, Unit of Physiotherapy, Institute of Neuroscience and Physiology, Sahlgrenska Academy, University of Gothenburg, , Gothenburg, Sweden
Locations (1):
- Närhälsan FaR-teamet centrala och västra Göteborg, Gothenburg, Region Västra Götaland, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blair SN. Physical inactivity: the biggest public health problem of the 21st century. Br J Sports Med. 2009 Jan;43(1):1-2. No abstract available. PMID 19136507
- [Background] Caspersen CJ, Powell KE, Christenson GM. Physical activity, exercise, and physical fitness: definitions and distinctions for health-related research. Public Health Rep. 1985 Mar-Apr;100(2):126-31. PMID 3920711
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1423-34. doi: 10.1249/mss.0b013e3180616b27. PMID 17762377
- [Background] Pavey TG, Taylor AH, Fox KR, Hillsdon M, Anokye N, Campbell JL, Foster C, Green C, Moxham T, Mutrie N, Searle J, Trueman P, Taylor RS. Effect of exercise referral schemes in primary care on physical activity and improving health outcomes: systematic review and meta-analysis. BMJ. 2011 Nov 4;343:d6462. doi: 10.1136/bmj.d6462. PMID 22058134
- [Background] Orrow G, Kinmonth AL, Sanderson S, Sutton S. Effectiveness of physical activity promotion based in primary care: systematic review and meta-analysis of randomised controlled trials. BMJ. 2012 Mar 26;344:e1389. doi: 10.1136/bmj.e1389. PMID 22451477
- [Background] Hallal PC, Lee IM. Prescription of physical activity: an undervalued intervention. Lancet. 2013 Feb 2;381(9864):356-7. doi: 10.1016/S0140-6736(12)61804-2. Epub 2012 Nov 28. No abstract available. PMID 23199848
- [Background] Kallings LV, Sierra Johnson J, Fisher RM, Faire Ud, Stahle A, Hemmingsson E, Hellenius ML. Beneficial effects of individualized physical activity on prescription on body composition and cardiometabolic risk factors: results from a randomized controlled trial. Eur J Cardiovasc Prev Rehabil. 2009 Feb;16(1):80-4. doi: 10.1097/HJR.0b013e32831e953a. PMID 19237997
- [Background] Leijon ME, Bendtsen P, Nilsen P, Festin K, Stahle A. Does a physical activity referral scheme improve the physical activity among routine primary health care patients? Scand J Med Sci Sports. 2009 Oct;19(5):627-36. doi: 10.1111/j.1600-0838.2008.00820.x. Epub 2008 Jul 8. PMID 18627557
- [Background] Olsson SJ, Borjesson M, Ekblom-Bak E, Hemmingsson E, Hellenius ML, Kallings LV. Effects of the Swedish physical activity on prescription model on health-related quality of life in overweight older adults: a randomised controlled trial. BMC Public Health. 2015 Jul 21;15:687. doi: 10.1186/s12889-015-2036-3. PMID 26193882
- [Background] Persson G, Ovhed I, Hansson EE. Simplified routines in prescribing physical activity can increase the amount of prescriptions by doctors, more than economic incentives only: an observational intervention study. BMC Res Notes. 2010 Nov 15;3:304. doi: 10.1186/1756-0500-3-304. PMID 21078135
- [Background] Sallis R, Franklin B, Joy L, Ross R, Sabgir D, Stone J. Strategies for promoting physical activity in clinical practice. Prog Cardiovasc Dis. 2015 Jan-Feb;57(4):375-86. doi: 10.1016/j.pcad.2014.10.003. Epub 2014 Oct 22. PMID 25459975
- [Background] Prochaska JO, DiClemente CC, Norcross JC. In search of how people change. Applications to addictive behaviors. Am Psychol. 1992 Sep;47(9):1102-14. doi: 10.1037//0003-066x.47.9.1102. PMID 1329589
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Grimby G, Borjesson M, Jonsdottir IH, Schnohr P, Thelle DS, Saltin B. The "Saltin-Grimby Physical Activity Level Scale" and its application to health research. Scand J Med Sci Sports. 2015 Dec;25 Suppl 4:119-25. doi: 10.1111/sms.12611. PMID 26589125
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] Sullivan M, Karlsson J, Ware JE Jr. The Swedish SF-36 Health Survey--I. Evaluation of data quality, scaling assumptions, reliability and construct validity across general populations in Sweden. Soc Sci Med. 1995 Nov;41(10):1349-58. doi: 10.1016/0277-9536(95)00125-q. PMID 8560302
- [Background] Grimby G. Physical activity and muscle training in the elderly. Acta Med Scand Suppl. 1986;711:233-7. doi: 10.1111/j.0954-6820.1986.tb08956.x. PMID 3535411
- [Derived] Ryen L, Lundqvist S, Cider A, Borjesson M, Larsson MEH, Hagberg L. Cost-Effectiveness of Prolonged Physical Activity on Prescription in Previously Non-Complying Patients: Impact of Physical Activity Mediators. Int J Environ Res Public Health. 2023 Feb 21;20(5):3801. doi: 10.3390/ijerph20053801. PMID 36900811
- [Derived] Lundqvist S, Borjesson M, Cider A, Hagberg L, Ottehall CB, Sjostrom J, Larsson MEH. Long-term physical activity on prescription intervention for patients with insufficient physical activity level-a randomized controlled trial. Trials. 2020 Sep 15;21(1):793. doi: 10.1186/s13063-020-04727-y. PMID 32933577